CLINICAL TRIAL: NCT04661566
Title: Optimizing a Multi-Modal Intervention to Reduce Health-Risking Sexual Behaviors: Component Selection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: USUHS.2020-055
Record Dates: First submitted 2020-10-23; First posted 2020-12-10 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Sexually Transmitted Infections; Pregnancy, Unplanned; Military Personnel
Keywords: Women's Health; Sexual and Reproductive Health; Military; Multiphase Optimization Strategy
MeSH Terms: conditions — Sexually Transmitted Diseases; Coitus | interventions — Educational Status; Risk

STUDY DESIGN:
Intervention Model Description: The MOST framework will be used. This study follows the optimization phase of the MOST framework where component selection experiments are conducted to experimentally evaluate the effectiveness of individual intervention components. Using a factorial design in this phase allows the effect of each intervention component to be evaluated and for observation of interaction effects while maximizing statistical power using a smaller sample size compared to an randomized controlled trial (RCT) powered similarly to explore individual components of an intervention. The optimization phase then allows for time and resources to be saved by ensuring only optimized components are retained after the RCT in the final intervention package.
Who Masked: Participant
Masking Description: Participants will not know the exact intervention conditions (i.e., what all of the intervention components are and what all of the possible combinations of intervention components there are)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (32):
- Education+Narratives+Skills+Scenarios+Future+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives, Skills, Scenarios, Future, and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Interactive Scenarios ("Scenarios"); Behavioral: Future Life Planning Tool ("Future"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Narratives+Skills+Scenarios+Future (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives, Skills, Scenarios, and Future
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Interactive Scenarios ("Scenarios"); Behavioral: Future Life Planning Tool ("Future")
- Education+Narratives+Skills+Scenarios+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives, Skills, Scenarios, and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Interactive Scenarios ("Scenarios"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Narratives+Skills+Scenarios (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives, Skills, and Scenarios
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Interactive Scenarios ("Scenarios")
- Education+Narratives+Skills+Future+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives, Skills, Future, and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Future Life Planning Tool ("Future"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Narratives+Skills+Future (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives, Skills, and Future
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Future Life Planning Tool ("Future")
- Education+Narratives+Skills+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives, Skills, and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Narratives+Skills (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives and Skills
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Skills Building Videos ("Skills")
- Education+Narratives+Scenarios+Future+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives. Scenarios, Future, and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Interactive Scenarios ("Scenarios"); Behavioral: Future Life Planning Tool ("Future"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Narratives+Scenarios+Future (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives, Scenarios, and Future
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Interactive Scenarios ("Scenarios"); Behavioral: Future Life Planning Tool ("Future")
- Education+Narratives+Scenarios+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives, Scenarios, and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Interactive Scenarios ("Scenarios"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Narratives+Scenarios (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives and Scenarios
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Interactive Scenarios ("Scenarios")
- Education+Narratives+Future+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives, Future, and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Future Life Planning Tool ("Future"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Narratives+Future (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives and Future
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Future Life Planning Tool ("Future")
- Education+Narratives+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Narratives (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Narratives
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Narrative Videos ("Narratives")
- Education+Skills+Scenarios+Future+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Skills, Scenarios, Future, and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Interactive Scenarios ("Scenarios"); Behavioral: Future Life Planning Tool ("Future"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Skills+Scenarios+Future (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Skills, Scenarios, and Future
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Interactive Scenarios ("Scenarios"); Behavioral: Future Life Planning Tool ("Future")
- Education+Skills+Scenarios+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Skills, Scenarios, and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Interactive Scenarios ("Scenarios"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Skills+Scenarios (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Skills and Scenarios
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Interactive Scenarios ("Scenarios")
- Education+Skills+Future+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Skills, Future, and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Future Life Planning Tool ("Future"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Skills+Future (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Skills Future
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Future Life Planning Tool ("Future")
- Education+Skills+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Skills and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Skills Building Videos ("Skills"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Skills (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Skills
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Skills Building Videos ("Skills")
- Education+Scenarios+Future+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Scenarios, Future, and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Interactive Scenarios ("Scenarios"); Behavioral: Future Life Planning Tool ("Future"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Scenarios+Future (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Scenarios and Future
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Interactive Scenarios ("Scenarios"); Behavioral: Future Life Planning Tool ("Future")
- Education+Scenarios+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Scenarios and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Interactive Scenarios ("Scenarios"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Scenarios (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Scenarios
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Interactive Scenarios ("Scenarios")
- Education+Future+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Future and Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Future Life Planning Tool ("Future"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education+Future (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Future
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Future Life Planning Tool ("Future")
- Education+Risk (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that includes the static educational component and the following components:
  Risk
  Interventions: Behavioral: Basic Education ("Education"); Behavioral: Epidemiological Risk Scenario ("Risk")
- Education (Experimental): Participants will receive a version of the Mission Wellness app (intervention) that only includes the static educational component.
  Interventions: Behavioral: Basic Education ("Education")

INTERVENTIONS:
Behavioral: Basic Education ("Education") — All participants will receive the basic educational component in the Mission Wellness app. This component will contain text and media (e.g., images, videos) to teach basic SRH topics. The exact information in this component will be determined by an assessment of baseline SRH knowledge at the start of the intervention.
Behavioral: Narrative Videos ("Narratives") — The narrative video component is a motivation-based component that includes stories of individuals engaging in positive and negative SRH behaviors that lead to either positive or negative outcomes, respectively, in a video format.
  Arms: Education+Narratives; Education+Narratives+Future; Education+Narratives+Future+Risk; Education+Narratives+Risk; Education+Narratives+Scenarios; Education+Narratives+Scenarios+Future; Education+Narratives+Scenarios+Future+Risk; Education+Narratives+Scenarios+Risk; Education+Narratives+Skills; Education+Narratives+Skills+Future; Education+Narratives+Skills+Future+Risk; Education+Narratives+Skills+Risk; Education+Narratives+Skills+Scenarios; Education+Narratives+Skills+Scenarios+Future; Education+Narratives+Skills+Scenarios+Future+Risk; Education+Narratives+Skills+Scenarios+Risk
Behavioral: Skills Building Videos ("Skills") — The skills-building videos component is a component rooted in behavioral skills that involves the provision of information on how to perform or engage positive SRH behaviors (e.g., correctly using a condom, what to expect when having a Pap smear) via instructional videos.
  Arms: Education+Narratives+Skills; Education+Narratives+Skills+Future; Education+Narratives+Skills+Future+Risk; Education+Narratives+Skills+Risk; Education+Narratives+Skills+Scenarios; Education+Narratives+Skills+Scenarios+Future; Education+Narratives+Skills+Scenarios+Future+Risk; Education+Narratives+Skills+Scenarios+Risk; Education+Skills; Education+Skills+Future; Education+Skills+Future+Risk; Education+Skills+Risk; Education+Skills+Scenarios; Education+Skills+Scenarios+Future; Education+Skills+Scenarios+Future+Risk; Education+Skills+Scenarios+Risk
Behavioral: Interactive Scenarios ("Scenarios") — The interactive scenarios are a behavioral skills-building component that walks through conversations surrounding SRH with select individuals (e.g., partner, healthcare provider), providing suggestions on how to have these conversations and why these conversations are important to have.
  Arms: Education+Narratives+Scenarios; Education+Narratives+Scenarios+Future; Education+Narratives+Scenarios+Future+Risk; Education+Narratives+Scenarios+Risk; Education+Narratives+Skills+Scenarios; Education+Narratives+Skills+Scenarios+Future; Education+Narratives+Skills+Scenarios+Future+Risk; Education+Narratives+Skills+Scenarios+Risk; Education+Scenarios; Education+Scenarios+Future; Education+Scenarios+Future+Risk; Education+Scenarios+Risk; Education+Skills+Scenarios; Education+Skills+Scenarios+Future; Education+Skills+Scenarios+Future+Risk; Education+Skills+Scenarios+Risk
Behavioral: Future Life Planning Tool ("Future") — The future life planning tool is a motivation-based component contains a series of questions to help users plan future goals to put current decision making related to SRH into perspective and provide suggestions on how to stay healthy now to be able to achieve those goals later.
  Arms: Education+Future; Education+Future+Risk; Education+Narratives+Future; Education+Narratives+Future+Risk; Education+Narratives+Scenarios+Future; Education+Narratives+Scenarios+Future+Risk; Education+Narratives+Skills+Future; Education+Narratives+Skills+Future+Risk; Education+Narratives+Skills+Scenarios+Future; Education+Narratives+Skills+Scenarios+Future+Risk; Education+Scenarios+Future; Education+Scenarios+Future+Risk; Education+Skills+Future; Education+Skills+Future+Risk; Education+Skills+Scenarios+Future; Education+Skills+Scenarios+Future+Risk
Behavioral: Epidemiological Risk Scenario ("Risk") — The risk component is an information- and motivation-based component with tailored epidemiological risk information about relative risk of contracting a specific STI and/or having an unintended pregnancy. Relative risk information will be determined by adjusting variables within the component (e.g., number of partners within the last month, percent of time using condoms).
  Arms: Education+Future+Risk; Education+Narratives+Future+Risk; Education+Narratives+Risk; Education+Narratives+Scenarios+Future+Risk; Education+Narratives+Scenarios+Risk; Education+Narratives+Skills+Future+Risk; Education+Narratives+Skills+Risk; Education+Narratives+Skills+Scenarios+Future+Risk; Education+Narratives+Skills+Scenarios+Risk; Education+Risk; Education+Scenarios+Future+Risk; Education+Scenarios+Risk; Education+Skills+Future+Risk; Education+Skills+Risk; Education+Skills+Scenarios+Future+Risk; Education+Skills+Scenarios+Risk

SUMMARY:
The goal of this project is to evaluate the components of the app-based intervention Mission Wellness to reduce health-risking sexual behaviors (HRSBs; e.g., condom non-use, multiple sexual partners) in active-duty members of the US Military to improve their sexual and reproductive health (SRH) and readiness to serve. Following the multiphase optimization strategy (MOST) framework, factorial component selection experiments (CSEs) will be conducted to evaluate which five experimental intervention components (i.e., Narratives, Skills, Scenarios, Future, and Risk) elicit the greatest improvements in the outcomes of interest given key constraints.

DETAILED DESCRIPTION:
Negative SRH outcomes (e.g., sexually transmitted infections [STIs], unintended pregnancy, STI-related cancers) reduce human performance and undermine military readiness. Service members face unique challenges to maintaining SRH during their military service. HRSBs (e.g., multiple sexual partners, unprotected sexual behavior) offer potential intervention targets to improve SRH. Electronic-health interventions are cost-effective and dynamic, and have the potential to reach millions of users as part of an overall strategy for individual behavior and systems change. In civilian populations, e-health interventions have demonstrated success in reducing HRSBs. However, effective HRSB-prevention interventions must consider the specific values, mission, and context of military populations and settings. The MOST framework is used to develop highly effective, efficient, and economic behavioral interventions that is particularly well suited to be used in this context.

This project aims to address this problem by delivering an optimized app-based prevention intervention package ready for evaluation via a subsequent randomized controlled trial (RCT). The specific purpose of this project is to determine which component(s) should be included in the packaged app-based intervention Mission Wellness for US service members based on their effects on the outcomes of interest (i.e., improved knowledge, motivation, and behavior skills related to SRH and reduced HRSBs) in no more than 25 minutes of content. The components tested in the factorial CSEs include: Narratives; Skills; Scenarios; Future; and Risk. Each component has two levels: "on" (included) or "off" (not included). Main and interaction effects of components will be measured to determine the components constituting the packaged intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 17 or older,
2. currently serving as active duty in the US military, and
3. willing to participate in all study activities if eligible and enrolled

Exclusion Criteria:

1. Does not meet eligibility criteria,
2. unable to read, speak, or comprehend English, or
3. unable or unwilling to give informed consent

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Change in SRH knowledge as assessed by measures of STI Knowledge | Baseline, within 3 weeks post-intervention, and 30-to-90 days post-intervention
  Change in SRH knowledge as assessed by STI Knowledge (Outcome 1) and Pregnancy and Birth Control Knowledge (Outcome 2).
  STI knowledge is measured on a dichotomous (true/false [outcome varies by item]) scale adapted from measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits and Gold's (1997) CD-ROM Technology to Increase Appropriate Self-Care and Preventive Behaviors among Army and Navy Women.
Change in SRH knowledge as assessed by measures of Pregnancy and Birth Control Knowledge | Baseline, within 3 weeks post-intervention, and 30-to-90 days post-intervention
  Change in SRH knowledge as assessed by STI Knowledge (Outcome 1) and Pregnancy and Birth Control Knowledge (Outcome 2).
  Pregnancy and Birth Control is measured on a dichotomous (true/false [outcome varies by item]) scale adapted from measures used in Frost's et al (2012) Young Adults' Contraceptive Knowledge, Norms, and Attitudes: Associations with Risk of Unintended Pregnancy and Gold's (1997) CD-ROM Technology to Increase Appropriate Self-Care and Preventive Behaviors among Army and Navy Women.
Change in perceived risk of having a negative SRH outcome as assessed by measures of Perceived Risk | Baseline, within 3 weeks post-intervention, and 30-to-90 days post-intervention
  Change in perceived risk of having a negative SRH outcome assessed by Perceived Risk on an 5-point ordinal scale (from "no risk" [better outcome] to "very high risk" [worse outcome]) adapted from measures used in Gold's (1997) CD-ROM Technology to Increase Appropriate Self-Care and Preventive Behaviors among Army and Navy Women.
Change in attitudes about SRH as assessed by measures of Condom Attitudes on a likert scale | Baseline, within 3 weeks post-intervention, and 30-to-90 days post-intervention
  Change in attitudes about SRH assessed by the composite Condom Attitudes (Outcome 4 and Outcome 5), composite Birth Control Attitudes (Outcome 6 and Outcome 7), and Norms (Outcome 8).
  Condom Attitudes is a composite score of Outcome 5 and a 7-point likert scale (from "strongly disagree" [1] to "strongly agree" [7; outcome varies by item]) adapted from Crosby's et al (2008) Correct Condom Use Self-Efficacy Scale (CCUSS) and Helweg-Larson and Collins' (1994) UCLA Multidimensional Condom Attitudes Scale (MCAS).
Change in attitudes about SRH as assessed by measures of Condom Attitudes on an ordinal item | Baseline, within 3 weeks post-intervention, and 30-to-90 days post-intervention
  Change in attitudes about SRH assessed by the composite Condom Attitudes (Outcome 4 and Outcome 5), composite Birth Control Attitudes (Outcome 6 and Outcome 7), and Norms (Outcome 8).
  Condom Attitudes is a composite score of Outcome 4 and a 5-point ordinal item (from "very positive" [better outcome] to "very negative" [worse outcome]) adapted from measures used in Gold's (1997) CD-ROM Technology to Increase Appropriate Self-Care and Preventive Behaviors among Army and Navy Women.
Change in attitudes about SRH as assessed by measures of Birth Control Attitudes on a likert-type scale | Baseline, within 3 weeks post-intervention, and 30-to-90 days post-intervention
  Change in attitudes about SRH assessed by the composite Condom Attitudes (Outcome 4 and Outcome 5), composite Birth Control Attitudes (Outcome 6 and Outcome 7), and Norms (Outcome 8).
  Birth Control Attitudes is a composite score of Outcome 7 and a 5-point likert-type scale (from "very positive" [better outcome] to "very negative" [worse outcome]) adapted from measures used in Gold's (1997) CD-ROM Technology to Increase Appropriate Self-Care and Preventive Behaviors among Army and Navy Women.
Change in attitudes about SRH as assessed by measures of Birth Control Attitudes on a likert scale | Baseline, within 3 weeks post-intervention, and 30-to-90 days post-intervention
  Change in attitudes about SRH assessed by the composite Condom Attitudes (Outcome 4 and Outcome 5), composite Birth Control Attitudes (Outcome 6 and Outcome 7), and Norms (Outcome 8).
  Birth Control Attitudes is a composite score of Outcome 6 and a 5-point likert scale (from "strongly agree" [1; worse outcome] to "strongly disagree" [5; better outcome]) adapted from measures used in Guzza and Hayford's (2018) Adolescent Reproductive and Contraceptive Knowledge and Attitudes and Adult Contraceptive Behavior.
Change in attitudes about SRH as assessed by measures of Norms | Baseline, within 3 weeks post-intervention, and 30-to-90 days post-intervention
  Change in attitudes about SRH assessed by the composite Condom Attitudes (Outcome 4 and Outcome 5), composite Birth Control Attitudes (Outcome 6 and Outcome 7), and Norms (Outcome 8).
  Change in attitudes about SRH assessed by Norms on a 5-point likert scale (from "strongly agree" to "strongly disagree" [no better/worse outcome]) adapted from measures used in Gold's (1997) CD-ROM Technology to Increase Appropriate Self-Care and Preventive Behaviors among Army and Navy Women.
Change in self-efficacy about SRH as assessed by measures of Condom/Birth Control Use | Baseline, within 3 weeks post-intervention, and 30-to-90 days post-intervention
  Change in self-efficacy about SRH assessed by Condom/Birth Control Use (Outcome 9) and Partner Communication/Negotiation (Outcome 10).
  Change in self-efficacy about SRH assessed by Condom/Birth Control Use on 5-point likert-type scales (from "not at all confident" [1; worse outcome] to "extremely confident" [5; better outcome]) adapted from Crosby's et al (2008) Correct Condom Use Self-Efficacy Scale (CCUSS) and Marin's et al (1997) Condom Self-Efficacy.
Change in self-efficacy about SRH as assessed by measures of Partner Communication/Negotiation | Baseline, within 3 weeks post-intervention, and 30-to-90 days post-intervention
  Change in self-efficacy about SRH assessed by Condom/Birth Control Use (Outcome 9) and Partner Communication/Negotiation (Outcome 10).
  Change in self-efficacy about SRH assessed by Partner Communication/Negotiation on a 4-point likert-type scale (from "very difficult" [1; worse outcome] to "very easy" [4; better outcome]) adapted from Noar's et al (2002) Condom Influence Strategy Questionnaire and Quinn-Nilas' et al (2016) Sexual Communication Self-Efficacy Scale.
Change in self-reported sexual behavior as assessed by measures of Sexual Behavior on ordinal items | Baseline and 30-to-90 days post-intervention
  Change in sexual behavior assessed by composite Sexual Behavior score (Outcomes 11-16).
  Sexual Behavior is a composite score of Outcomes 12-16 and ordinal (from "never" [worse outcome] to "all the time" [better outcome]) items adapted from measures used in Booth-Kewley's et al (2001) One-Year Follow-Up Evaluation of the Sexually Transmitted Disease/Human Immunodeficiency Virus Intervention Program in a Marine Corps sample.
Change in self-reported sexual behavior as assessed by measures of Sexual Behavior on yes/no/dont-know items | Baseline and 30-to-90 days post-intervention
  Change in sexual behavior assessed by composite Sexual Behavior score (Outcomes 11-16).
  Sexual Behavior is a composite score of Outcomes 11 and 13-16, and yes/no/dont-know (nominal; outcome varies by item) items adapted from measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits, Hwang's et al (2007) Sexual Behaviors After Universal Screening of Sexually Transmitted Infections in Healthy Young Women, and Booth-Kewley's et al (2001) One-Year Follow-Up Evaluation of the Sexually Transmitted Disease/Human Immunodeficiency Virus Intervention Program in a Marine Corps sample.
Change in self-reported sexual behavior as assessed by measures of Sexual Behavior on no/yes,previously/yes,currently items | Baseline and 30-to-90 days post-intervention
  Change in sexual behavior assessed by composite Sexual Behavior score (Outcomes 11-16).
  Sexual Behavior is a composite score of Outcomes 11-12 and 14-16 and no/yes,previously/yes,currently (nominal; no better/worse outcome) items adapted from measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits, Hwang's et al (2007) Sexual Behaviors After Universal Screening of Sexually Transmitted Infections in Healthy Young Women, and Booth-Kewley's et al (2001) One-Year Follow-Up Evaluation of the Sexually Transmitted Disease/Human Immunodeficiency Virus Intervention Program in a Marine Corps sample.
Change in self-reported sexual behavior as assessed by measures of Sexual Behavior on dichotomous items | Baseline and 30-to-90 days post-intervention
  Change in sexual behavior assessed by composite Sexual Behavior score (Outcomes 11-16).
  Sexual Behavior is a composite score of Outcomes 11-13 and 15-16 and dichotomous (yes/no [outcome varies by item]) items adapted from measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits, Hwang's et al (2007) Sexual Behaviors After Universal Screening of Sexually Transmitted Infections in Healthy Young Women, and Booth-Kewley's et al (2001) One-Year Follow-Up Evaluation of the Sexually Transmitted Disease/Human Immunodeficiency Virus Intervention Program in a Marine Corps sample.
Change in self-reported sexual behavior as assessed by measures of Sexual Behavior on open response (number input) items | Baseline and 30-to-90 days post-intervention
  Change in sexual behavior assessed by composite Sexual Behavior score (Outcomes 11-16).
  Sexual Behavior is a composite score of Outcomes 11-14 and 16 and open response (number input) items adapted from measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits, Hwang's et al (2007) Sexual Behaviors After Universal Screening of Sexually Transmitted Infections in Healthy Young Women, and Booth-Kewley's et al (2001) One-Year Follow-Up Evaluation of the Sexually Transmitted Disease/Human Immunodeficiency Virus Intervention Program in a Marine Corps sample.
Change in self-reported sexual behavior as assessed by measures of Sexual Behavior on nominal items | Baseline and 30-to-90 days post-intervention
  Change in sexual behavior assessed by composite Sexual Behavior score (Outcomes 11-16).
  Sexual Behavior is a composite score of Outcomes 11-15 and nominal items (main/casual other [no better/worse outcome]) adapted from measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits, Hwang's et al (2007) Sexual Behaviors After Universal Screening of Sexually Transmitted Infections in Healthy Young Women, and Booth-Kewley's et al (2001) One-Year Follow-Up Evaluation of the Sexually Transmitted Disease/Human Immunodeficiency Virus Intervention Program in a Marine Corps sample.
Change in self-reported sexual behavior as assessed by measures of Sexual Behavioral Intentions on ordinal items | Within 3 weeks post-intervention
  Change in sexual behavior assessed by composite Sexual Behavioral Intentions (Outcomes 17-21).
  Sexual Behavior Intentions is a composite score of Outcomes 18-21 and 5-point ordinal (from "never" [worse outcome] to "all of the time" [better outcome]) items adapted from measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits, Hwang's et al (2007) Sexual Behaviors After Universal Screening of Sexually Transmitted Infections in Healthy Young Women, and Booth-Kewley's et al (2001) One-Year Follow-Up Evaluation of the Sexually Transmitted Disease/Human Immunodeficiency Virus Intervention Program in a Marine Corps sample.
Change in self-reported sexual behavior as assessed by measures of Sexual Behavioral Intentions on yes/no/dont-know items | Within 3 weeks post-intervention
  Change in sexual behavior assessed by composite Sexual Behavioral Intentions (Outcomes 17-21).
  Sexual Behavior Intentions is a composite score of Outcomes 17 and 19-21 and nominal (yes/no/dont-know [outcome varies by item]) items adapted from measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits, Hwang's et al (2007) Sexual Behaviors After Universal Screening of Sexually Transmitted Infections in Healthy Young Women, and Booth-Kewley's et al (2001) One-Year Follow-Up Evaluation of the Sexually Transmitted Disease/Human Immunodeficiency Virus Intervention Program in a Marine Corps sample.
Change in self-reported sexual behavior as assessed by measures of Sexual Behavioral Intentions on dichotomous items | Within 3 weeks post-intervention
  Change in sexual behavior assessed by composite Sexual Behavioral Intentions (Outcomes 17-21).
  Sexual Behavior Intentions is a composite score of Outcomes 17-18 and 20-21 and dichotomous (yes/no [outcome varies by item]) items adapted from measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits, Hwang's et al (2007) Sexual Behaviors After Universal Screening of Sexually Transmitted Infections in Healthy Young Women, and Booth-Kewley's et al (2001) One-Year Follow-Up Evaluation of the Sexually Transmitted Disease/Human Immunodeficiency Virus Intervention Program in a Marine Corps sample.
Change in self-reported sexual behavior as assessed by measures of Sexual Behavioral Intentions on open response (number input) items | Within 3 weeks post-intervention
  Change in sexual behavior assessed by composite Sexual Behavioral Intentions (Outcomes 17-21).
  Sexual Behavior Intentions is a composite score of Outcomes 17-19 and 21 and open response (number input) items adapted from measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits, Hwang's et al (2007) Sexual Behaviors After Universal Screening of Sexually Transmitted Infections in Healthy Young Women, and Booth-Kewley's et al (2001) One-Year Follow-Up Evaluation of the Sexually Transmitted Disease/Human Immunodeficiency Virus Intervention Program in a Marine Corps sample.
Change in self-reported sexual behavior as assessed by measures of Sexual Behavioral Intentions | Within 3 weeks post-intervention
  Change in sexual behavior assessed by composite Sexual Behavioral Intentions (Outcomes 17-21).
  Sexual Behavior Intentions is a composite score of Outcomes 17-20 and a 7-point likert-type (from "definitely" [better outcome] to "not likely at all" [worse outcome]) scale adapted from measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits, Hwang's et al (2007) Sexual Behaviors After Universal Screening of Sexually Transmitted Infections in Healthy Young Women, and Booth-Kewley's et al (2001) One-Year Follow-Up Evaluation of the Sexually Transmitted Disease/Human Immunodeficiency Virus Intervention Program in a Marine Corps sample.
Quality and satisfaction of healthcare experiences as assessed by measures of Health Care on ordinal items (from "very helpful" to "not helpful at all") | Baseline and 30-to-90 days post-intervention
  Quality and satisfaction of healthcare experiences assessed by composite Health Care (Outcomes 22-27).
  Health Care is a composite score of Outcomes 23-27 and on 5-point ordinal or likert-type (from "very helpful" [better outcome] to "not helpful at all" [worse outcome]) items adapted from measures used in Gold's (1997) CD-ROM Technology to Increase Appropriate Self-Care and Preventive Behaviors among Army and Navy Women.
Quality and satisfaction of healthcare experiences as assessed by measures of Health Care on ordinal items (from "strongly agree" to "strongly disagree") | Baseline and 30-to-90 days post-intervention
  Quality and satisfaction of healthcare experiences assessed by composite Health Care (Outcomes 22-27).
  Health Care is a composite score of Outcomes 22 and 24-27 and on 5-point ordinal or likert-type (from "strongly agree" [better outcome] to "strongly disagree" [worse outcome]) items adapted from measures used in Gold's (1997) CD-ROM Technology to Increase Appropriate Self-Care and Preventive Behaviors among Army and Navy Women.
Quality and satisfaction of healthcare experiences as assessed by measures of Health Care on ordinal items (from "to much" to "some to little") | Baseline and 30-to-90 days post-intervention
  Quality and satisfaction of healthcare experiences assessed by composite Health Care (Outcomes 22-27).
  Health Care is a composite score of Outcomes 22-23 and 25-27 and on 5-point ordinal or likert-type (from "too much" to "some too little" [no better/worse outcome]) items adapted from measures used in Gold's (1997) CD-ROM Technology to Increase Appropriate Self-Care and Preventive Behaviors among Army and Navy Women.
Quality and satisfaction of healthcare experiences as assessed by measures of Health Care on yes/no/dont-know nominal items | Baseline and 30-to-90 days post-intervention
  Quality and satisfaction of healthcare experiences assessed by composite Health Care (Outcomes 22-27).
  Health Care is a composite score of Outcomes 22-24 and 26-27 and yes/no/dont-know (no better/worse outcome) items adapted from measures used in Gold's (1997) CD-ROM Technology to Increase Appropriate Self-Care and Preventive Behaviors among Army and Navy Women.
Quality and satisfaction of healthcare experiences as assessed by measures of Health Care on no/yes,recent/yes,not-recent nominal items | Baseline and 30-to-90 days post-intervention
  Quality and satisfaction of healthcare experiences assessed by composite Health Care (Outcomes 22-27).
  Health Care is a composite score of Outcomes 22-25 and 27 and no/yes,recent/yes,not-recent (no better/worse outcome) nominal items adapted from measures used in Gold's (1997) CD-ROM Technology to Increase Appropriate Self-Care and Preventive Behaviors among Army and Navy Women.
Quality and satisfaction of healthcare experiences as assessed by measures of Health Care on a cumulative scale | Baseline and 30-to-90 days post-intervention
  Quality and satisfaction of healthcare experiences assessed by composite Health Care (Outcomes 22-27).
  Health Care is a composite score of Outcomes 22 and 24-26 and a cumulative (outcome varies by item) scales adapted from measures used in Gold's (1997) CD-ROM Technology to Increase Appropriate Self-Care and Preventive Behaviors among Army and Navy Women.
Quality and satisfaction of healthcare provider interactions as assessed by measures of Patient-Provider Communication | Baseline
  Quality and satisfaction of healthcare provider interactions as assessed by Patient-Provider Communication on a 5-point likert-type scale (from "I do not agree" [worse outcome] to "I fully agree" [better outcome]) adapted from Bieber's et al (2010) Questionnaire on the Quality of Physician-Patient Interaction (QQPPI)
Change in self-reported mental health as assessed by Depression (PHQ-2) | Baseline and 30-to-90 days post-intervention
  Change in mental health assessed by Depression on the Patient Health Questionnaire-2 (PHQ-2) (from "not at all" [better outcome] to "nearly every day" [worse outcome])
Change in self-reported mental health as assessed by Anxiety (HAI) | Baseline and 30-to-90 days post-intervention
  Change in mental health assessed by the Anxiety on the Health Anxiety Inventory (HAI)
Intervention acceptability as assessed by measures on Acceptability | Within 3 weeks post-intervention
  Acceptability of the intervention assessed by composite measures on Acceptability (Outcomes 31-33).
  Acceptability is a composite score of Outcome 32-33 and a 5-point ordinal or likert-type scale (from "do not agree at all" [worse outcome] to "agree completely" [better outcome]) adapted from Stoyanov's et al (2015) Mobile App Rating Scale and measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits and Kelley's et al (2005) An Evaluation of a Sexual Assault Prevention and Advocacy Program for US Navy Personnel.
Intervention acceptability as assessed by measures on Acceptability as open-ended items | Within 3 weeks post-intervention
  Acceptability of the intervention assessed by composite measures on Acceptability (Outcomes 31-33).
  Acceptability is a composite score of Outcome 31 and 33 and open-ended items adapted from Stoyanov's et al (2015) Mobile App Rating Scale and measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits and Kelley's et al (2005) An Evaluation of a Sexual Assault Prevention and Advocacy Program for US Navy Personnel.
Intervention acceptability as assessed by measures on Acceptability on a rating scale | Within 3 weeks post-intervention
  Acceptability of the intervention assessed by composite measures on Acceptability (Outcomes 31-33).
  Acceptability is a composite score of Outcome 31-32 and a rating scale (from 1 ["not at all likely"; worse outcome] to 10 ["extremely likely"; better outcome]) adapted from Stoyanov's et al (2015) Mobile App Rating Scale and measures used in Acari's et al (2004) Feasibility and Short-Term Impact of Linked Education and Urine Screening Interventions for Chlamydia and Gonorrhea in Male Army Recruits and Kelley's et al (2005) An Evaluation of a Sexual Assault Prevention and Advocacy Program for US Navy Personnel.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan R Landoll, PhD, Principal Investigator — Uniformed Services University of the Health Sciences; Sara E Vargas, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Uniformed Services University of the Health Sciences, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT04661566/Prot_SAP_005.pdf
  • Informed Consent Form (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT04661566/ICF_004.pdf